CLINICAL TRIAL: NCT04067050
Title: A Clinical Study of the Biofinity Energys Soft Contact Lens in Users of Digital Devices
Brief Title: A Clinical Study of the Comfilcon A Asphere Soft Contact Lens in Users of Digital Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EX-MKTG-105
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Ametropia
MeSH Terms: conditions — Refractive Errors | interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- comfilcon A asphere (Experimental): Subjects will wear their comfilcon A asphere contact lenses for two months. Lenses will be worn on a daily wear, reusable basis for at least 8 hours per day, 5 days per week.
  Interventions: Device: comfilcon A asphere
- Habitual Spectacles (Active Comparator): Subjects will wear their single vision habitual spectacles for two months for at least 8 hours per day, 5 days per week.
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: comfilcon A asphere — Contact Lens
  Other Names: test
  Arms: comfilcon A asphere
Device: Spectacles — Habitual spectacles
  Other Names: Control; Single Vision Spectacles
  Arms: Habitual Spectacles

SUMMARY:
The aim of this work is to investigate the clinical performance and subjective acceptance of the comfilcon A asphere contact lens when compared to single-vision spectacles in subjects who have never worn contact lenses and who use digital devices (such as phones, tablets, laptops, desktop computers) for at least 4 hours per day on at least 5 days per week.

DETAILED DESCRIPTION:
The aim of this clinical work is to compare the clinical performance and subjective acceptance of comfilcon A asphere contact lens when compared to single-vision spectacles in subjects who use digital devices (phones, tablets, laptops, desktop computers) for at least 4 hours per day on at least 5 days per week. Subjects will be randomized to use either their habitual spectacles or the study contact lenses for two months.

ELIGIBILITY:
Inclusion Criteria:

* They are between 18 and 35 years of age (inclusive).
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They are a 'neophyte' (i.e. someone who has not worn contact lenses previously, with the exception for the purposes of a trial fitting, lasting up to one week).
* They have a contact lens spherical prescription between -1.00 to -6.25D (inclusive) based on the ocular refraction.
* They have a cylindrical correction of -0.875DC or less in each eye based on the ocular refraction
* They own and habitually wear single vision spectacles used for both distance and near vision, including computer and digital device use.
* Their single vision spectacles have a mean sphere equivalent within ±0.50D of that of the refraction found in the study for each eye (after having taken lens effectivity into account).
* They are willing to be fitted with contact lenses and understand they may be randomized to either group.
* They are willing to wear the contact lenses (if relevant) or spectacles for at least 8 hours per day, 5 days per week.
* They typically use digital devices for a minimum of 4 hours per day, 5 days per week.
* They agree not to change the spectacles they will wear for digital device use for the duration of the study.
* They agree not to participate in other clinical research for the duration of the study.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops (including comfort drops) or ointment on a regular basis.
* The spectacles they use for digital device viewing on the study have been made with specialist features for computer use, digital eye fatigue or are multifocal/bifocal.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or breastfeeding.
* They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
* They have evidence of a heterotropia or decompensating heterotropia on cover test.
* They have a history of having been prescribed prism in their spectacles (by self report).
* They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: One Month
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Started | 32 | 29
Completed | 28 | 29
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 4 | 0
Period: Two Month
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Started | 22 (6 subjects discontinued after 1 month visit. 22 Subjects continued the study.) | 29
Completed | 20 | 29
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Comfilcon A Asphere: Subjects were randomized to use the study contact lenses for two months.
- Habitual Spectacles: Subjects were randomized to wear habitual spectacles for two months.
- Total: Total of all reporting groups
Arm/Group | Comfilcon A Asphere | Habitual Spectacles | Total
Number analyzed (Participants) | 32 | 29 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 29 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (3.9) | 22.9 (4.4) | 23.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 29 | 61

OUTCOME MEASURES:

1. Primary Outcome: Symptom of Burning
Description: Symptom of burning measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of burning was measured only for subjects who had frequency of symptom of burning on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.16 (0.37) | 0.21 (0.49)
  Intensity: number analyzed (Participants) | 6 | 5
  Intensity | 1.00 (0.00) | 1.00 (0.00)

2. Primary Outcome: Symptom of Burning
Description: as for outcome 1
Time Frame: 1 month
Population: One subject scores was not measured for Habitual spectacles group. Intensity of symptom of burning was measured only for subjects who had frequency of symptom of burning on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.11 (0.31) | 0.29 (0.53)
  Intensity: number analyzed (Participants) | 3 | 7
  Intensity | 1.00 (0.00) | 1.14 (0.38)

3. Primary Outcome: Symptom of Burning
Description: as for outcome 1
Time Frame: 2 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.00 (0.00) | 0.17 (0.38)
  Intensity: number analyzed (Participants) | 0 | 5
  Intensity |  | 1.00 (0.00)

4. Primary Outcome: Symptom of Itching
Description: Symptom of itching measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of itching was measured only for subjects who had frequency of itching on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.41 (0.56) | 0.52 (0.57)
  Intensity: number analyzed (Participants) | 12 | 14
  Intensity | 1.08 (0.29) | 1.00 (0.00)

5. Primary Outcome: Symptom of Itching
Description: as for outcome 4
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of itching was measured only for subjects who had frequency of itching on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.68 (0.55) | 0.36 (0.56)
  Intensity: number analyzed (Participants) | 18 | 9
  Intensity | 1.00 (0.00) | 1.00 (0.00)

6. Primary Outcome: Symptom of Itching
Description: as for outcome 4
Time Frame: Two Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.45 (0.51) | 0.41 (0.50)
  Intensity: number analyzed (Participants) | 9 | 29
  Intensity | 1.00 (0.00) | 1.00 (0.00)

7. Primary Outcome: Symptom of Feeling of Foreign Body
Description: Symptom of feeling of foreign body measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of feeling of foreign body was measured only for subjects who had frequency of feeling of foreign body on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.19 (0.40) | 0.17 (0.38)
  Intensity: number analyzed (Participants) | 6 | 5
  Intensity | 1.33 (0.52) | 1.20 (0.45)

8. Primary Outcome: Symptom of Feeling of Foreign Body
Description: as for outcome 7
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of feeling of foreign body was measured only for subjects who had frequency of feeling of foreign body on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.75 (0.59) | 0.11 (0.31)
  Intensity: number analyzed (Participants) | 19 | 3
  Intensity | 1.00 (0.00) | 1.00 (0.00)

9. Primary Outcome: Symptom of Feeling of Foreign Body
Description: as for outcome 7
Time Frame: Two Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.50 (0.61) | 0.21 (0.41)
  Intensity: number analyzed (Participants) | 9 | 6
  Intensity | 1.00 (0.00) | 1.00 (0.00)

10. Primary Outcome: Symptom of Tearing
Description: Symptom of tearing measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of tearing was measured only for subjects who had frequency of symptom of tearing on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.53 (0.51) | 0.43 (0.63)
  Intensity: number analyzed (Participants) | 17 | 11
  Intensity | 1.06 (0.24) | 1.18 (0.40)

11. Primary Outcome: Symptom of Tearing
Description: as for outcome 10
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of tearing was measured only for subjects who had frequency of symptom of tearing on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.39 (0.57) | 0.33 (0.48)
  Intensity: number analyzed (Participants) | 10 | 10
  Intensity | 1.00 (0.00) | 1.10 (0.32)

12. Primary Outcome: Symptom of Tearing
Description: as for outcome 10
Time Frame: Two Months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.35 (0.49) | 0.45 (0.57)
  Intensity: number analyzed (Participants) | 7 | 12
  Intensity | 1.00 (0.00) | 1.08 (0.29)

13. Primary Outcome: Symptom of Excessive Blinking
Description: Symptom of excessive blinking measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of excessive blinking was measured only for subjects who had frequency of symptom of excessive blinking on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.25 (0.51) | 0.38 (0.56)
  Intensity: number analyzed (Participants) | 8 | 10
  Intensity | 1.00 (0.00) | 1.10 (0.32)

14. Primary Outcome: Symptom of Excessive Blinking
Description: as for outcome 13
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of excessive blinking was measured only for subjects who had frequency of symptom of excessive blinking on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.46 (0.51) | 0.29 (0.53)
  Intensity: number analyzed (Participants) | 13 | 7
  Intensity | 1.00 (0.00) | 1.14 (0.38)

15. Primary Outcome: Symptom of Excessive Blinking
Description: as for outcome 13
Time Frame: Two Months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.35 (0.49) | 0.17 (0.38)
  Intensity: number analyzed (Participants) | 7 | 5
  Intensity | 1.00 (0.00) | 1.20 (0.45)

16. Primary Outcome: Symptom of Eye Redness
Description: Symptom of eye redness measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of eye redness was measured only for subjects who had frequency of symptom of eye redness on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.28 (0.46) | 0.21 (0.41)
  Intensity: number analyzed (Participants) | 9 | 6
  Intensity | 1.11 (0.33) | 1.00 (0.00)

17. Primary Outcome: Symptom of Eye Redness
Description: as for outcome 16
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of eye redness was measured only for subjects who had frequency of symptom of eye redness on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.36 (0.56) | 0.18 (0.39)
  Intensity: number analyzed (Participants) | 9 | 5
  Intensity | 1.00 (0.00) | 1.00 (0.00)

18. Primary Outcome: Symptom of Eye Redness
Description: as for outcome 16
Time Frame: Two Months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.20 (0.41) | 0.24 (0.44)
  Intensity: number analyzed (Participants) | 4 | 7
  Intensity | 1.00 (0.00) | 1.00 (0.00)

19. Primary Outcome: Symptom of Eye Pain
Description: Symptom of eye pain measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of eye pain was measured only for subjects who had frequency of symptom of eye pain on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.34 (0.55) | 0.34 (0.61)
  Intensity: number analyzed (Participants) | 10 | 8
  Intensity | 1.10 (0.32) | 1.13 (0.35)

20. Primary Outcome: Symptom of Eye Pain
Description: as for outcome 19
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of eye pain was measured only for subjects who had frequency of symptom of eye pain on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.14 (0.36) | 0.25 (0.44)
  Intensity: number analyzed (Participants) | 4 | 7
  Intensity | 1.00 (0.00) | 1.00 (0.00)

21. Primary Outcome: Symptom of Eye Pain
Description: as for outcome 19
Time Frame: Two Months
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.00 (0.00) | 0.31 (0.54)
  Intensity: number analyzed (Participants) | 0 | 8
  Intensity |  | 1.00 (0.00)

22. Primary Outcome: Symptom of Heavy Eyelids
Description: Symptom of heavy eyelids measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of heavy eyelids was measured only for subjects who had frequency of symptom of heavy eyelids on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.56 (0.62) | 0.45 (0.51)
  Intensity: number analyzed (Participants) | 16 | 13
  Intensity | 1.13 (0.34) | 1.00 (0.00)

23. Primary Outcome: Symptom of Heavy Eyelids
Description: as for outcome 22
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of heavy eyelids was measured only for subjects who had frequency of symptom of heavy eyelids on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.39 (0.50) | 0.46 (0.58)
  Intensity: number analyzed (Participants) | 11 | 12
  Intensity | 1.00 (0.00) | 1.17 (0.39)

24. Primary Outcome: Symptom of Heavy Eyelids
Description: as for outcome 22
Time Frame: Two Months
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.35 (0.49) | 0.48 (0.63)
  Intensity: number analyzed (Participants) | 6 | 12
  Intensity | 1.00 (0.00) | 1.08 (0.29)

25. Primary Outcome: Symptom of Dryness
Description: Symptom of dryness measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of dryness was measured only for subjects who had frequency of symptom of dryness on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.38 (0.55) | 0.48 (0.51)
  Intensity: number analyzed (Participants) | 11 | 14
  Intensity | 1.18 (0.40) | 1.00 (0.00)

26. Primary Outcome: Symptom of Dryness
Description: as for outcome 25
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of dryness was measured only for subjects who had frequency of symptom of dryness on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.75 (0.70) | 0.43 (0.50)
  Intensity: number analyzed (Participants) | 17 | 12
  Intensity | 1.06 (0.24) | 1.00 (0.00)

27. Primary Outcome: Symptom of Dryness
Description: as for outcome 25
Time Frame: Two Months
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.75 (0.55) | 0.48 (0.57)
  Intensity: number analyzed (Participants) | 14 | 13
  Intensity | 1.07 (0.27) | 1.15 (0.38)

28. Primary Outcome: Symptom of Blurred Vision
Description: Symptom of blurred vision measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of blurred vision was measured only for subjects who had frequency of symptom of blurred vision on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.34 (0.48) | 0.45 (0.51)
  Intensity: number analyzed (Participants) | 12 | 13
  Intensity | 1.00 (0.00) | 1.00 (0.00)

29. Primary Outcome: Symptom of Blurred Vision
Description: as for outcome 28
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of blurred vision was measured only for subjects who had frequency of symptom of blurred vision on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.54 (0.58) | 0.25 (0.44)
  Intensity: number analyzed (Participants) | 14 | 7
  Intensity | 1.00 (0.00) | 1.14 (0.38)

30. Primary Outcome: Symptom of Blurred Vision
Description: as for outcome 28
Time Frame: Two Months
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.35 (0.49) | 0.28 (0.45)
  Intensity: number analyzed (Participants) | 7 | 8
  Intensity | 1.00 (0.00) | 1.00 (0.00)

31. Primary Outcome: Symptom of Double Vision
Description: Symptom of double vision measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of double vision was measured only for subjects who had frequency of symptom of double vision on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.06 (0.25) | 0.07 (0.37)
  Intensity: number analyzed (Participants) | 3 | 1
  Intensity | 1.00 (0.00) | 1.00 (0.00)

32. Primary Outcome: Symptom of Double Vision
Description: as for outcome 31
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of double vision was measured only for subjects who had frequency of symptom of double vision on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.11 (0.31) | 0.07 (0.26)
  Intensity: number analyzed (Participants) | 3 | 2
  Intensity | 1.00 (0.00) | 1.00 (0.00)

33. Primary Outcome: Symptom of Double Vision
Description: as for outcome 31
Time Frame: Two Months
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.05 (0.22) | 0.07 (0.26)
  Intensity: number analyzed (Participants) | 1 | 2
  Intensity | 1.00 (0.00) | 1.00 (0.00)

34. Primary Outcome: Symptom of Difficulty Focusing For Near Vision
Description: Symptom of difficulty focusing for near vision measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of difficulty focusing for near vision was measured only for subjects who had frequency of symptom of difficulty focusing for near vision on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.28 (0.46) | 0.41 (0.57)
  Intensity: number analyzed (Participants) | 10 | 11
  Intensity | 1.10 (0.32) | 1.00 (0.00)

35. Primary Outcome: Symptom of Difficulty Focusing For Near Vision
Description: as for outcome 34
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of difficulty focusing for near vision was measured only for subjects who had frequency of symptom of difficulty focusing for near vision on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.18 (0.39) | 0.29 (0.46)
  Intensity: number analyzed (Participants) | 5 | 8
  Intensity | 1.00 (0.00) | 1.00 (0.00)

36. Primary Outcome: Symptom of Difficulty Focusing For Near Vision
Description: as for outcome 34
Time Frame: Two Months
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.45 (0.51) | 0.14 (0.35)
  Intensity: number analyzed (Participants) | 9 | 4
  Intensity | 1.00 (0.00) | 1.00 (0.00)

37. Primary Outcome: Symptom of Increased Sensitivity to Light
Description: Symptom of increased sensitivity to light measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of increased sensitivity to light was measured only for subjects who had frequency of symptom of increased sensitivity to light on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.59 (0.67) | 0.48 (0.63)
  Intensity: number analyzed (Participants) | 16 | 12
  Intensity | 1.19 (0.40) | 1.17 (0.39)

38. Primary Outcome: Symptom of Increased Sensitivity to Light
Description: as for outcome 37
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of increased sensitivity to light was measured only for subjects who had frequency of symptom of increased sensitivity to light on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.25 (0.44) | 0.36 (0.62)
  Intensity: number analyzed (Participants) | 7 | 8
  Intensity | 1.00 (0.00) | 1.13 (0.35)

39. Primary Outcome: Symptom of Increased Sensitivity to Light
Description: as for outcome 37
Time Frame: Two Months
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.10 (0.31) | 0.24 (0.44)
  Intensity: number analyzed (Participants) | 1 | 7
  Intensity | 1.00 (0.00) | 1.14 (0.38)

40. Primary Outcome: Symptom of Colored Haloes Around Objects
Description: Symptom of colored haloes around objects measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of colored haloes around objects was measured only for subjects who had frequency of symptom of colored haloes around objects on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.16 (0.45) | 0.17 (0.47)
  Intensity: number analyzed (Participants) | 4 | 4
  Intensity | 1.25 (0.50) | 1.00 (0.00)

41. Primary Outcome: Symptom of Colored Haloes Around Objects
Description: as for outcome 40
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of colored haloes around objects was measured only for subjects who had frequency of symptom of colored haloes around objects on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.11 (0.31) | 0.07 (0.26)
  Intensity: number analyzed (Participants) | 3 | 2
  Intensity | 1.00 (0.00) | 1.00 (0.00)

42. Primary Outcome: Symptom of Colored Halos Around Objects
Description: Symptom of colored halos around objects measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Two Months
Population: as for outcome 40
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.10 (0.31) | 0.07 (0.26)
  Intensity: number analyzed (Participants) | 2 | 2
  Intensity | 1.00 (0.00) | 1.00 (0.00)

43. Primary Outcome: Symptom of Feeling That Sight is Worsening
Description: Symptom of feeling that sight is worsening measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of feeling that sight is worsening was measured only for subjects who had frequency of symptom of feeling that sight is worsening on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 28
units on a scale
  Frequency | 0.34 (0.60) | 0.48 (0.51)
  Intensity: number analyzed (Participants) | 9 | 14
  Intensity | 1.00 (0.00) | 1.07 (0.27)

44. Primary Outcome: Symptom of Feeling That Sight is Worsening
Description: as for outcome 43
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of feeling that sight is worsening was measured only for subjects who had frequency of symptom of feeling that sight is worsening on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.25 (0.44) | 0.36 (0.49)
  Intensity: number analyzed (Participants) | 7 | 10
  Intensity | 1.00 (0.00) | 1.10 (0.32)

45. Primary Outcome: Symptom of Feeling That Sight is Worsening
Description: as for outcome 43
Time Frame: Two Months
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.20 (0.41) | 0.45 (0.63)
  Intensity: number analyzed (Participants) | 4 | 11
  Intensity | 1.00 (0.00) | 1.00 (0.00)

46. Primary Outcome: Symptom of Headache
Description: Symptom of headache measured by frequency on a scale of 0-2 (0-never, 1- occasionally, 2- often/always) and intensity on a scale of 1-2 (1- moderate 2- intense).
Time Frame: Baseline
Population: Intensity of symptom of headache was measured only for subjects who had frequency of symptom of headache on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 32 | 29
units on a scale
  Frequency | 0.72 (0.63) | 0.69 (0.60)
  Intensity: number analyzed (Participants) | 21 | 18
  Intensity | 1.10 (0.30) | 1.06 (0.24)

47. Primary Outcome: Symptom of Headache
Description: as for outcome 46
Time Frame: One Month
Population: One subject score was not measured for Habitual spectacles group. Intensity of symptom of headache was measured only for subjects who had frequency of symptom of headache on a scale of 1 - occasionally and 2- often/always
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 28 | 28
units on a scale
  Frequency | 0.33 (0.48) | 0.54 (0.58)
  Intensity: number analyzed (Participants) | 9 | 14
  Intensity | 1.22 (0.44) | 1.14 (0.36)

48. Primary Outcome: Symptom of Headache
Description: as for outcome 46
Time Frame: Two Months
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
Number analyzed (Participants) | 20 | 29
units on a scale
  Frequency | 0.30 (0.47) | 0.55 (0.51)
  ntensity: number analyzed (Participants) | 6 | 16
  ntensity | 1.00 (0.00) | 1.13 (0.34)

ADVERSE EVENTS:
Time Frame: From baseline visit up to two months, a total of two months.
Arm/Group | Comfilcon A Asphere | Habitual Spectacles
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 1/32 | 0/29
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comfilcon A Asphere (N=32) | Habitual Spectacles (N=29)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT04067050/Prot_SAP_000.pdf